CLINICAL TRIAL: NCT05433740
Title: Comparison of Two Different Methods for ProsealTM Laryngeal Mask Fixation
Brief Title: LMA Fixation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, expert doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 04.04.2022 134/13
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Fixation Device; Complications
Keywords: laryngeal mask airway; fixation; fiberoptic bronchoscope

STUDY DESIGN:
Intervention Model Description: Group I: Adjustable ligament or Group II, adhesive tape
Who Masked: Participant
Masking Description: undergoing urologic surgery using LMA with ASA Physical Status I-III, Mallampati score I-II, and >18 years of age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Adjustable ligament (Experimental): In the adjustable ligament method, binding tape with a button at one end and button holes along the band was wrapped around the outer end of the bite-block section of the device. The ends of the tape were then passed over the outer end of the bite block between two tubes and adjusted at or above the ear level (except neck veins), and fixed by inserting the button through the appropriate hole.
  Interventions: Device: Proseal Laryngeal mask fixation
- Group II: Adhesive tape (No Intervention): The laryngeal mask was fixed using the standard method using adhesive tape.

INTERVENTIONS:
Device: Proseal Laryngeal mask fixation — fixation with Proseal Laryngeal mask adjustable ligament
  Arms: Group I: Adjustable ligament

SUMMARY:
Proseal laryngeal mask airway (LMA) is frequently used for safe airway management in modern anesthesia. Improper fixation of the LMA may result in subsequent displacement despite initial correct placement. In this study, researchers aimed to present the detection method researchers developed for PLMA, which is different from the classical methods.

PLMA will place with a new fixation method in adult patients in the lithotomy position who will undergo uretero-renoscopic lithotripsy. The fixation will prepare by sewing a button on one end of the adjustable elastic. Successful insertion will assess clinically (capnogram, appropriate chest excursion, and the absence of an audible leak at a peak inspiratory pressure of 20 cm H2O) and with a fiberoptic bronchoscope (FOB) (grade and distance visible to vocal cords). At the end of the operation, it will be examined whether there is any displacement.

SPSS 21.0 (Version 22.0, SPSS, Inc, Chicago, IL, USA) program will be used for statistical analysis. After applying the Shapiro-Wilk test for normality, the student's t test will be used if the distribution is normal, and the Mann-Whitey U test will be used if the distribution is not normal. Fisher's exact test or chi-square test will be used for categorical variables. Results p<0.05 will be considered significant.

DETAILED DESCRIPTION:
Proseal laryngeal mask airway (LMA) is frequently used for safe airway management in modern anesthesia. Improper fixation of the LMA may result in subsequent displacement despite initial correct placement. In this study, researchers aimed to present the detection method researchers developed for PLMA, which is different from the classical methods.

PLMA will place with a new fixation method in adult patients in the lithotomy position who will undergo uretero-renoscopic lithotripsy. The fixation will prepare by sewing a button on one end of the adjustable elastic. Successful insertion will assess clinically (capnogram, appropriate chest excursion, and the absence of an audible leak at a peak inspiratory pressure of 20 cm H2O) and with a fiberoptic bronchoscope (FOB) (grade and distance visible to vocal cords). At the end of the operation, it will be examined whether there is any displacement.

SPSS 21.0 (Version 22.0, SPSS, Inc, Chicago, IL, USA) program will be used for statistical analysis. After applying the Shapiro-Wilk test for normality, the student's t test will be used if the distribution is normal, and the Mann-Whitey U test will be used if the distribution is not normal. Fisher's exact test or chi-square test will be used for categorical variables. Results p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing urologic surgery using LMA
* ASA Physical Status I-III
* Mallampati score I-II

  * 18 years

Exclusion Criteria:

* Patients who did not want to participate in the study
* Restricted mouth opening
* BMI ≥ 35 kg/m2
* Risk of airway malformation and aspiration (gastroesophageal reflux, hiatal hernia, history of previous gastric surgery, GIS motility disorder)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
laryngeal mask correct insertion and than fixation | intraoperative period (From the insertion of the laryngeal mask airway to its removal at the end of the procedure)
  The placement and fixation of the laryngeal mask will be evaluated by measuring the end-tidal carbon dioxide value with the aid of a capnogram, the formation of appropriate chest extension, and the absence of audible leakage at 20 cm H2O peak inspiratory pressure.

SECONDARY OUTCOMES:
Evaluation of successful laryngeal mask placement with a fiberoptic bronchoscope (FOB) | intraoperative period (From the insertion of the laryngeal mask airway to its removal at the end of the procedure)
  To evaluate the best fiberoptic bronchoscopic view while insertion of proseal laryngeal mask

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Science, Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chandan SN, Sharma SM, Raveendra US, Rajendra Prasad B. Fiberoptic assessment of laryngeal mask airway placement: a comparison of blind insertion and insertion with the use of a laryngoscope. J Maxillofac Oral Surg. 2009 Jun;8(2):95-8. doi: 10.1007/s12663-009-0025-8. Epub 2009 Aug 11. PMID 23139483
- [Result] Garc'a-Aguado R. Fixation of the ProSeal Laryngeal Mask Airway with a gauze bandage. Anaesthesia. 2005 Jul;60(7):726. doi: 10.1111/j.1365-2044.2005.04277.x. No abstract available. PMID 15960739
- [Result] Cook TM, Lee G, Nolan JP. The ProSeal laryngeal mask airway: a review of the literature. Can J Anaesth. 2005 Aug-Sep;52(7):739-60. doi: 10.1007/BF03016565. PMID 16103390